CLINICAL TRIAL: NCT07021820
Title: Multispectral Optoacoustic Tomography for Advanced Imaging of Centronuclear Myopathy
Acronym: MOSAIC
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, Study Chair, University of Erlangen-Nürnberg Medical School
Other Study IDs: 25-120-Bm
Record Dates: First submitted 2025-05-15; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Centronuclear Myopathy
Keywords: MSOT; centronuclear myopathy; MOSAIC
MeSH Terms: conditions — Myopathies, Structural, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CNM: patients with diagnosed centronuclear myopathy
  Interventions: Diagnostic Test: MSOT
- HV: Healthy control
  Interventions: Diagnostic Test: MSOT

INTERVENTIONS:
Diagnostic Test: MSOT — Multispectral optoacoustic tomography (MSOT) enables the detection of specific endogenous chromophores such as collagen, myoglobin or haemoglobin using a non-invasive approach comparable to conventional ultrasound. Instead of sound waves, MSOT illuminates the tissue with near-infrared light of transient energy, which is absorbed and leads to thermoelastic expansion of certain molecules. This expansion generates ultrasound waves that are detected by the same device. The multispectral illumination and unmixing then enable the precise localization and quantification of muscle-specific subcellular structures. MSOT has already shown the potential to visualize the muscle structure and clinical extent of muscle disease in patients with Duchenne muscular dystrophy, spinal muscular atrophy and the late-onset Pompe disease (LOPD) and to distinguish these patients from healthy volunteers. To date, there is no optoacoustic data on CNM.

SUMMARY:
Twenty patients with centronuclear myopathy and twenty age- and sex-matched, muscle-healthy controls will undergo diagnostic examination. Study participants will undergo physical examination, clinical and functional testing, and multispectral optoacoustic tomography (MSOT) scanning at predefined muscle sites (paraspinal muscles, trapezius muscle, deltoid muscle, forearm flexors, quadriceps muscle, adductor muscles, ischiocrural muscles, triceps surae muscle, and tibialis anterior).

DETAILED DESCRIPTION:
Centronuclear myopathy (CNM) belongs to the group of congenital myopathies. These are named after their histopathological feature: the nucleus is localized in the center of the muscle cell instead of its physiological position at the periphery. CNM is so rare that there are only epidemiological data available for the group of congenital myopathies as a whole. The incidence is estimated at 0.06 per 1,000 live births.

CNM is genetically and clinically heterogeneous. Identified gene mutations affect proteins involved in membrane remodeling, transport, and excitation-contraction coupling.

Patients with CNM usually present with muscle weakness and hypotonia in early childhood. The severity of the disease varies depending on the underlying genotype and ranges from reduced exercise tolerance and ptosis to floppy infant syndrome and respiratory failure. One example of a very severe course is the X-linked form caused by a Myotubularin 1 (MTM1) nonsense mutation (XL-MTM). Affected patients become symptomatic in the neonatal period and usually die in childhood or adolescence. In contrast, patients with the Dynamin 2 (DNM2) mutation have a later onset and milder disease progression. In the few reported patients with Bridging Integrator 1 (BIN1) mutations, onset occurs in infancy or adulthood with a moderate disease course. Ryanodine receptor 1 (RYR1)-associated CNMs also vary in terms of age of onset and disease severity.

Diagnosis is based on molecular genetic testing and muscle biopsy. However, these techniques are not widely available, are time-consuming, and invasive. Anesthesia is usually required for young patients.

Multispectral optoacoustic tomography (MSOT) enables the detection of specific endogenous chromophores such as collagen, myoglobin, or hemoglobin using a non-invasive approach comparable to conventional ultrasound. Instead of sound waves, MSOT uses near-infrared light pulses that are absorbed by tissue, causing thermoelastic expansion of certain molecules. This expansion generates ultrasound waves, which are then detected by the same device. The multispectral illumination and signal unmixing enable precise localization and quantification of muscle-specific subcellular structures. MSOT has already demonstrated the potential to visualize muscle structure and disease extent in patients with Duchenne muscular dystrophy, spinal muscular atrophy, and late-onset Pompe disease (LOPD), and to distinguish these patients from healthy volunteers. To date, there are no optoacoustic data available for CNM.

The aim of this study is to gain molecular insights into muscle degeneration in CNM patients for the first time. To develop a comprehensive picture of the optoacoustic characteristics of CNM, patients of different ages and disease severities will be recruited. Due to the rarity and small number of CNM cases, recruitment is challenging. Therefore, the opportunity should be taken to offer study participation to as many patients as possible at the patient meeting in Bad Nauheim from May 29 to June 1, 2025. In addition to non-invasive, radiation-free imaging, clinical-functional tests will be conducted as part of the study. These include muscle strength testing (MRC score) and the timed "get up and go" test. Various accessible muscle groups will be scanned using MSOT, including the paraspinal muscles and trapezius muscle, as well as the following limb muscles on both sides: deltoid, biceps brachii, forearm flexors, quadriceps femoris, adductors, hamstrings (ischiocrural muscles), triceps surae, and tibialis anterior.

ELIGIBILITY:
CNM arm:

Inclusion Criteria: diagnosed CNM; minimum of 2 years of age

Exclusion Criteria:

* Pregnancy
* Nursing mothers
* Tattoo in the area of the examination field
* Subcutaneous fatty tissue > 3 cm

HV:

Inclusion criteria: minimum of 2 years of age

Exclusion criteria:

* any signs/history of muscle diseases
* Pregnancy
* Nursing mothers
* Tattoo in the area of the examination field
* Subcutaneous fatty tissue > 3 cm

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: n= 20 CNM n = 20 HV
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Optoacoustic spectrum of MSOT Imaging (all in arbitrary units) | Day 1
  Comparison of optoacoustic spectrum from patients with diagnosed CNM and their age- and sex matched Healthy Volunteers

SECONDARY OUTCOMES:
Comparison of MSOT-Derived Hemoglobin and Myoglobin Signals | Day 1
  Quantitative comparison of MSOT-derived hemoglobin and myoglobin signals (arbitrary units).
Comparison of Oxygenated vs. Deoxygenated Hemoglobin Signal | Day 1
  Quantitative comparison of oxygenated and deoxygenated hemoglobin signals.
Comparison of Oxygenated Hemoglobin and Lipid Signal | Day 1
  Quantitative comparison of oxygenated hemoglobin and lipid signals.
Comparison of deoxygenated Hemoglobin and Lipid Signal | Day 1
  Quantitative comparison of deoxygenated hemoglobin and lipid signals.
Comparison of oxygenated Hemoglobin and Collagen Signal | Day 1
  Quantitative comparison of oxygenated hemoglobin and collagen signals.
Comparison of deoxygenated Hemoglobin and Collagen Signal | Day 1
  Quantitative comparison of deoxygenated hemoglobin and collagen signals.
Comparison of Lipid and Collagen Signal | Day 1
  Quantitative comparison of Lipid and collagen signals.
Comparison of Lipid and Myoglobin Signal | Day 1
  Quantitative comparison of Lipid and Myoglobin signals.
Comparison of Collagen and Myoglobin Signal | Day 1
  Quantitative comparison of Collagen and Myoglobin signals.
Correlation of Hemoglobin Signal with Disease Duration and Patient Age | Day 1
  Unit of Measure: Correlation coefficient (Pearson's r or Spearman's ρ)
Correlation of Myoglobin Signal with Disease Duration and Patient Age | Day 1
  Unit of Measure: Correlation coefficient (Pearson's r or Spearman's ρ)
Correlation of oxygenated and deoxygenated Hemoglobin Signal with Disease Duration and Patient Age | Day 1
  Unit of Measure: Correlation coefficient (Pearson's r or Spearman's ρ)
Correlation of Lipid Signal with Disease Duration and Patient Age | Day 1
  Unit of Measure: Correlation coefficient (Pearson's r or Spearman's ρ)
Correlation of Collagen Signal with Disease Duration and Patient Age | Day 1
  Unit of Measure: Correlation coefficient (Pearson's r or Spearman's ρ)
Correlation of Hemoglobin Signal with MRC Muscle Strength | Day 1
  Unit of Measure: Correlation coefficient (MRC scale: ordinal, 1-5)
Correlation of Myoglobin Signal with MRC Muscle Strength | Day 1
  Unit of Measure: Correlation coefficient (MRC scale: ordinal, 1-5)
Correlation of oxygenated and dexoygenated Hemoglobin with MRC Muscle Strength | Day 1
  Unit of Measure: Correlation coefficient (MRC scale: ordinal, 1-5)
Correlation of Lipid Signal with MRC Muscle Strength | Day 1
  Unit of Measure: Correlation coefficient (MRC scale: ordinal, 1-5)
Correlation of Collagen Signal with MRC Muscle Strength | Day 1
  Unit of Measure: Correlation coefficient (MRC scale: ordinal, 1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, PD Dr. med. habil. Dr. rer. b, Study Chair — Kinder- & Jugendklinik, Erlangen
Locations (1):
- Uniklinikum Erlangen, Erlangen, Bavaria, Germany

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT07021820/Prot_SAP_000.pdf